CLINICAL TRIAL: NCT01936883
Title: IMPROVING QUALITY OF LIFE AFTER OPTIMAL RADIOTHERAPY FOR INTERMEDIATE AND HIGH RISK PROSTATE CANCER: A Randomized Comparison of HDR Versus LDR BRACHYTHERAPY BOOST
Brief Title: Improving Quality of Life After Prostate Brachytherapy: a Comparison of HDR and LDR Brachytherapy
Acronym: BrachyQOL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H13-02139
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: prostatic neoplasm; brachytherapy; quality of life; high dose rate; low dose rate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LDR boost (Active Comparator): After completion of 46 Gy of external beam radiotherapy subjects will undergo a permanent seed radioactive implant to the prostate using iodine-125 seeds to deliver a dose of 110 Gy
  Interventions: Radiation: LDR
- HDR boost (Active Comparator): Subjects in this arm will undergo an HDR implant to deliver 15 Gy to the prostate prior to commencing the external beam component of their treatment.
  Interventions: Radiation: HDR

INTERVENTIONS:
Radiation: HDR — High dose rate brachytherapy
  Arms: HDR boost
Radiation: LDR — Low dose rate brachytherapy boost
  Arms: LDR boost

SUMMARY:
Optimal non surgical treatment of prostate cancer requires dose escalation which is frequently provided by adding a brachytherapy "boost" to a short course of external beam radiotherapy. The hypothesis in this randomized study is that a High Dose Rate (HDR) brachytherapy boost leads to equivalent or better Prostate Specific Antigen (PSA) recurrence-free survival when compared to a Low Dose Rate (LDR) brachytherapy boost and that it is associated with a more favorable toxicity profile and improved quality of life.

DETAILED DESCRIPTION:
Men with intermediate or high risk prostate cancer who are technically suitable for prostate brachytherapy based on prostate size and voiding function and who are interested in this modality of treatment will be approached for randomization between either high dose rate (single 15 Gray) or low dose rate permanent seed implant (110 Gray) brachytherapy. Baseline International Prostate Symptom score, Quality of Life Assessment and International Index of Erectile Function will be recorded and then every 3 months for the first year and every 6 months to 3 years. Androgen deprivation treatment is allowed for 6 or 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Upper tier intermediate risk with at least 2 of the following factors

  1. Tumor-Nodes-Metastases Tumor stage T2B or greater
  2. Gleason Score 7
  3. PSA > 10
  4. > 50% of the biopsies positive
* OR High risk prostate cancer with one of the following factors

  1. T3a
  2. Gleason Score8-10
  3. PSA >20
* Positive prostate biopsy within 12 months (reviewed centrally)
* International Prostate Symptom Score < 16
* Prostate volume < 60 cc
* Negative staging CT and Bone scan within 3 months prior to registration
* History and physical examination within 90 days prior to registration
* European Cooperative Oncology Group performance status 0-1 prior to registration
* Age >45
* Patient suitable for procedure under anesthesia

Exclusion Criteria:

* Prior invasive malignancy (except non melanoma skin cancer) unless disease-free for at least 3 years prior to registration
* Previous prostatectomy, cryotherapy or High Intensity Focussed Ultrasound for prostate cancer
* Previous pelvic irradiation or prostate brachytherapy

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2014-01; Primary Completion 2019-12 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Compare Quality of Life between two arms as measured by EPIC questionnaire | 6 months
  Quality of life will be measured through validated instruments including International Prostate Symptom Score (IPSS), the International Index of Erectile Function ((IEF), and the urinary, bowel and sexual domains of the Expanded Prostate Cancer Index Composite (EPIC). IPSS has 7 questions related to voiding symptoms, each scored 0-5, with a higher score indicating worse symptoms. IIEF has 5 questions, each scored 0-5 with a higher score indicating better function. EPIC has several questions for each domain with an overall higher score associated with better QoL in that domain.

SECONDARY OUTCOMES:
Quality of Life long term | 5 years
  Quality of Life will be assessed to 5 years using the validated instruments International Prostate Symptom Score, International Index Erectile Function and EPIC

OTHER OUTCOMES:
Efficacy: cancer free status | 10 years
  regular PSA monitoring every 6 months to 3 years and then annually to determine PSA recurrence free survival

CONTACTS AND LOCATIONS:
Overall Officials: Juanita M Crook, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency Center for the Southern Interior, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bachand F, Martin AG, Beaulieu L, Harel F, Vigneault E. An eight-year experience of HDR brachytherapy boost for localized prostate cancer: biopsy and PSA outcome. Int J Radiat Oncol Biol Phys. 2009 Mar 1;73(3):679-84. doi: 10.1016/j.ijrobp.2008.05.003. Epub 2008 Oct 27. PMID 18963537
- [Background] Schmid M, Crook JM, Batchelar D, Araujo C, Petrik D, Kim D, Halperin R. A phantom study to assess accuracy of needle identification in real-time planning of ultrasound-guided high-dose-rate prostate implants. Brachytherapy. 2013 Jan-Feb;12(1):56-64. doi: 10.1016/j.brachy.2012.03.002. Epub 2012 Apr 17. PMID 22513104
- [Background] Morton GC, Loblaw DA, Chung H, Tsang G, Sankreacha R, Deabreu A, Zhang L, Mamedov A, Cheung P, Batchelar D, Danjoux C, Szumacher E. Health-related quality of life after single-fraction high-dose-rate brachytherapy and hypofractionated external beam radiotherapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2011 Aug 1;80(5):1299-305. doi: 10.1016/j.ijrobp.2010.04.046. Epub 2010 Aug 12. PMID 20708853
- [Background] Pieters BR, de Back DZ, Koning CC, Zwinderman AH. Comparison of three radiotherapy modalities on biochemical control and overall survival for the treatment of prostate cancer: a systematic review. Radiother Oncol. 2009 Nov;93(2):168-73. doi: 10.1016/j.radonc.2009.08.033. Epub 2009 Sep 11. PMID 19748692
- [Background] Deutsch I, Zelefsky MJ, Zhang Z, Mo Q, Zaider M, Cohen G, Cahlon O, Yamada Y. Comparison of PSA relapse-free survival in patients treated with ultra-high-dose IMRT versus combination HDR brachytherapy and IMRT. Brachytherapy. 2010 Oct-Dec;9(4):313-8. doi: 10.1016/j.brachy.2010.02.196. Epub 2010 Aug 4. PMID 20685176
- [Background] Stock RG, Stone NN, Cesaretti JA, Rosenstein BS. Biologically effective dose values for prostate brachytherapy: effects on PSA failure and posttreatment biopsy results. Int J Radiat Oncol Biol Phys. 2006 Feb 1;64(2):527-33. doi: 10.1016/j.ijrobp.2005.07.981. Epub 2005 Oct 19. PMID 16242258